CLINICAL TRIAL: NCT01281592
Title: Open-Label, Phase 1 Study of LOR-253 HCl in Patients With Advanced or Metastatic Solid Tumours
Brief Title: A Study of LOR-253 HCl in Patients With Advanced or Metastatic Solid Tumours
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aptose Biosciences Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 253-SOL1-01
Record Dates: First submitted 2011-01-20; First posted 2011-01-24 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2014-02

CONDITIONS: Advanced or Metastatic Solid Tumours

ARMS (1):
- LOR-253 HCl (Experimental): LOR-253 HCl will be given in ascending doses until the maximum administered dose or appropriate target dose is reached. A biomarker study of up to 10 patients will be conducted upon achieving appropriate dose level.
  Interventions: Drug: LOR-253 HCl

INTERVENTIONS:
Drug: LOR-253 HCl — LOR-253 HCl will be given in ascending doses starting from 20 mg/m2 until the maximum administered dose or appropriate target dose is reached. Patient will be treated on LOR-253 HCl for 2 cycles for the evaluation.
  Other Names: No other names are used.

SUMMARY:
This is an open-label, phase 1 study to determine the maximum tolerated dose (MTD) or appropriate target dose if MTD not reached to identify the recommended phase 2 dose of LOR-253 HCl in patients with advanced or metastatic solid tumours.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 18 years of age or older.
2. Histologically confirmed diagnosis of solid tumour for which no effective therapy is available or that is unresponsive to conventional therapy.
3. Meet laboratory parameter requirements at study entry.

Exclusion Criteria:

1. Chemotherapy, radiotherapy, biologic therapy, immunotherapy or any other investigational drugs within 21 days of beginning study treatment with LOR-253 HCl.
2. A hematologic malignancy.
3. A history of brain or other central nervous system metastases.
4. Have a presence of a significant infection.
5. Clinically significant autoimmune disease.
6. Uncontrolled intercurrent illness.
7. With iron or copper overload syndromes.
8. Pregnancy or breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2011-01; Primary Completion 2013-07 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose (MTD) or appropriate target dose if MTD not reached to identify the recommended phase 2 dose of LOR-253 HCl in patients with advanced or metastatic solid tumours. | 8 weeks

SECONDARY OUTCOMES:
To characterize the safety profile of LOR-253 HCl when administered to patients with advanced or metastatic solid tumours. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Cercek, M.D., Principal Investigator — Memorial Sloan Kettering Cancer Center; Jennifer Wheler, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - MD Anderson Cancer Center, Houston, Texas